CLINICAL TRIAL: NCT07142941
Title: Effects of Exercise and/or β-hydroxy-β-methylbutyrate Supplementation on Muscle Mass, Physical Performance and Insulin Resistance in Older Diabetes With Low Muscle Mass: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Exercise and/or HMB in Older Diabetes With Low Muscle Mass
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Shangling (Other)
Responsible Party: Sponsor-Investigator, Wu Shangling, Doctor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: exercise and/or HMB
Record Dates: First submitted 2025-07-25; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Diabetes; Low Muscle Mass
Keywords: low muscle mass; diabetes; HMB; exercise
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HMB + Exercise (Experimental): Participants were instructed to take active products including 3000 mg calcium-HMB per day, and allocated to the exercise programs were provided 45 min of supervised sessions on 2 nonconsecutive days per week
  Interventions: Dietary Supplement: HMB; Behavioral: Exercise
- Placebo + Exercise (Experimental): Participants allocated to the exercise programs were provided 45 min of supervised sessions on 2 nonconsecutive days per week, and were instructed to take active products including equal in quality resistant dextrin per day
  Interventions: Behavioral: Exercise; Dietary Supplement: Placebo
- HMB + Education (Experimental): Participants were instructed to take active products including 3000 mg calcium-HMB per day, and were given health education and educational manuals.
  Interventions: Dietary Supplement: HMB; Other: Education
- Placebo + Education (Placebo Comparator): Participants were instructed to take active products including equal in quality resistant dextrin per day, and were given health education and educational manuals
  Interventions: Dietary Supplement: Placebo; Other: Education

INTERVENTIONS:
Dietary Supplement: HMB — Participants were instructed to take active products including 3000 mg calcium-HMB per day
  Arms: HMB + Education; HMB + Exercise
Behavioral: Exercise — Participants allocated to the exercise programs were provided 45 min of supervised sessions on 2 nonconsecutive days per week
  Arms: HMB + Exercise; Placebo + Exercise
Dietary Supplement: Placebo — Participants were instructed to take active products including equal in quality resistant dextrin per day
  Arms: Placebo + Education; Placebo + Exercise
Other: Education — Participants were given health education and educational manuals
  Arms: HMB + Education; Placebo + Education

SUMMARY:
The investigators aimed to examine if β-hydroxy-β-methylbutyrate (HMB) supplementation enhances the effects of exercise on muscle mass, physical performance and insulin resistance and observe potential residual effects in older diabetes with low muscle mass, and to find the optimal treatment plan.

DETAILED DESCRIPTION:
The interaction between exercise and nutritional supplementation is unclear among older diabetes at risk of sarcopenia. The investigators aimed to examine if β-hydroxy-β-methylbutyrate (HMB) supplementation enhances the effects of exercise on muscle mass, physical performance and insulin resistance and observe potential residual effects in older diabetes with low muscle mass, and to find the optimal treatment plan. This 12-wk, randomized, double-blind, placebo controlled, 2 × 2 factorial design (exercise-only, HMB-only, both, and none) trial included 120 older diabetes aged 60-80 y with skeletal muscle index <5.7 kg/m2 for women, and <7.0 kg/m2 for men, and was followed by a 12-wk observational period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-80 ;
* Diagnosis of T2DM
* Low muscle mass: met a reference value for low muscle mass defined by the Asian Working Group for Sarcopenia (AWGS) criteria with skeletal muscle index <5.7 kg/m2 for women and <7.0 kg/m2 for men

Exclusion Criteria:

* Individuals who had an organic disease of the nervous system;
* Who were restricted from engaging in exercise by a medical doctor;
* Who was unconscious and unable to complete the questionnaire;
* Who used other supplementations for muscle mass gain;
* Who had impaired cardiac, kidney, or liver function.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
muscle mass | 0 and 12 weeks
  Body composition including muscle mass was measured using a segmental multifrequency bioelectrical impedance device (Inbody)
Handgrip strength | 0 and 12 weeks
  Handgrip strength was measured using a handheld Smedley-type dynamometer.
5-repetition sit-to-stand time | 0 and 12 weeks
  Participants folded their arms across their chests and were instructed to stand-up completely and make firm contact when sitting. Timing began on the command "go" and ceased when the participants sat after the fifth stand-up. Participants were allowed a practice trial of 2 repetitions before the timing of 2 test trials of 5 repetitions.

SECONDARY OUTCOMES:
insulin resistance index | 0 and 12 weeks
  Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) was calculated as follow:
  HOMA-IR=(Fasting Insulin (μU/mL)×Fasting Glucose (mg/dL))/405

CONTACTS AND LOCATIONS:
Overall Officials: Shangling Wu, Study Chair — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No